CLINICAL TRIAL: NCT03055585
Title: Applying Wolbachia to Eliminate Dengue (AWED): A Non-blinded Cluster Randomised Controlled Trial to Assess the Efficacy of Wolbachia-infected Mosquito Deployments to Reduce Dengue Incidence in Yogyakarta, Indonesia
Brief Title: Applying Wolbachia to Eliminate Dengue
Acronym: AWED
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Distancing and movement restrictions of the COVID-19 emergency response made continuation of clinic-based and field entomological trial activities infeasible
Sponsor: Gadjah Mada University (Other)
Collaborators: Monash University (Other); The Tahija Foundation (Unknown)
Responsible Party: Principal Investigator, Riris Andono Ahmad, Director of Center for Tropical Medicine, Faculty of Medicine, Universitas Gadjah Mada, Gadjah Mada University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UGM_KE/FK/105/EC
Record Dates: First submitted 2017-02-14; First posted 2017-02-16 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Dengue; Zika Virus Infection; Chikungunya Fever
Keywords: Wolbachia; Ae. aegypti; Indonesia; Dengue; Cluster-randomised trial
MeSH Terms: conditions — Dengue; Zika Virus Infection; Chikungunya Fever

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): Deployment of Wolbachia-infected Aedes aegypti mosquitoes
  Interventions: Biological: Wolbachia-infected Aedes aegypti mosquitoes; Other: standard practice dengue control
- Comparison arm (Other): Standard practice dengue control activities
  Interventions: Other: standard practice dengue control

INTERVENTIONS:
Biological: Wolbachia-infected Aedes aegypti mosquitoes — Deployment of Wolbachia-infected Aedes aegypti mosquitoes
  Arms: Intervention arm
Other: standard practice dengue control — standard practice dengue control activities conducted by dengue control program

SUMMARY:
This cluster randomised trial will evaluate the efficacy of Wolbachia-infected Aedes aegytpi mosquitoes in reducing dengue cases in Yogyakarta City, Indonesia

DETAILED DESCRIPTION:
Primary objective:

To assess the efficacy of community-based deployments of Wolbachia-infected Aedes aegypti mosquitoes in reducing the incidence of symptomatic, virologically-confirmed dengue cases of any severity in Yogyakarta residents aged 3-45 years in release areas, relative to non-release areas.

Secondary objectives:

* To measure the efficacy of the Wolbachia method against each of the four DENV serotypes.
* To measure the efficacy of the Wolbachia method in reducing the incidence of symptomatic virologically confirmed Zika virus and chikungunya virus infection in release areas, relative to non-release areas
* To quantify the level of human mobility within Yogyakarta City, and estimate the proportion of residents' exposure time that they spend outside the treatment arm to which they were randomised
* To determine whether community-based deployment of Wolbachia-infected Ae. aegypti mosquitoes reduces the abundance of wild-type Ae. aegypti adults, or alternatively, alters the abundance of adults from Aedes species other than Ae. aegypti (e.g. Ae. albopictus)

Study setting:

The study will be conducted in Yogyakarta City and Bantul District, both located in the province of Yogyakarta Special Region, Indonesia.The study site is 26 km2 in size, including 24 km2 within Yogyakarta City, and 2km2 in the adjacent Bantul District. The total population of the study area is approximately 350,000.

Study design:

A cluster randomised trial with a test-negative design will be conducted. The study site will be divided into 24 clusters. The intervention will be allocated using constrained block randomisation with a parallel 1:1 assignment of intervention and control.

The intervention is the deployment of Wolbachia-infected Aedes aegypti mosquitoes. Wolbachia deployments will be conducted in intervention clusters with the aim of achieving Wolbachia establishment (>80% mean Wolbachia prevalence in trapped mosquitoes) throughout intervention areas within one year.

The impact of Wolbachia deployments on dengue incidence will be assessed by comparing the exposure distribution (probability of living in a Wolbachia-treated area) among virologically-confirmed dengue cases presenting to a network of public primary clinics (Puskesmas), against the exposure distribution among patients with febrile illness of non-arboviral aetiology presenting to the same network of clinics in the same temporal windows. Dengue cases and arbovirus-negative controls will be sampled concurrently from within the population of patients presenting with febrile illness to the study clinic network, with case or control status classified retrospectively based on the results of laboratory diagnostic testing.

A re-estimation of sample size requirements was conducted in January 2019 after one year of recruitment. The initial power calculation used 1000 dengue cases and 4000 non-dengue controls allocated to each cluster based on historical proportions of dengue cases and other febrile illnesses, assuming no variation in the proportion of cases by cluster. This method was found to overestimate power for small samples by not taking into account randomness in the sampling. The sample size re-estimation included power estimates for 200, 400, 600, 800 and 1000 dengue cases with 4 times as many controls allocated to each cluster by sampling from a multinomial distribution, which incorporated added randomness by allowing the proportion of cases allocated to each cluster to vary across simulations. The re-estimation found that 400 dengue cases plus four times as many controls would be sufficient to detect a 50% reduction in dengue incidence with 80% power.

Participant selection:

Participants will be enrolled from within the population of patients presenting with undifferentiated fever of 1-4 days duration, to one of the participating local health clinics (Puskesmas).

All patients meeting the inclusion criteria will be invited to participate in the study. From baseline historical data we expect approximately 5000 participants per annum to be enrolled.

Enrolment will continue for up to 36 months.

Analysis plan:

Permutation tests and standard regression models will be used to estimate the relative risk of dengue in Wolbachia-treated versus untreated clusters, accounting for the non-independence of study participants resident in the same intervention cluster, and temporal matching of dengue cases and test-negative controls.

The intention-to-treat analysis will consider Wolbachia exposure as binary depending on the allocation of the cluster of residence.

The per-protocol analysis will consider Wolbachia exposure as a continuous weighted index based on Wolbachia prevalence in trapped mosquitoes in the cluster of residence, either with or without weighting for time spent in other clusters visited during the ten days prior to illness onset.

ELIGIBILITY:
Inclusion Criteria:

* Fever (either self-reported or objectively measured, e.g. (tympanic membrane temperature ≥38oC)) of 1-4 days duration, and where onset was prior to the day of presentation
* Aged between 3-45 years old
* Resided in the study area every night for the 10 days preceding illness onset

Exclusion Criteria:

* Localising features suggestive of a specific diagnosis other than an arboviral infection e.g. severe diarrhea, otitis, pneumonia
* Prior enrollment in the study within the previous 4 weeks

Ages: 3 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 8173 (Actual)
Dates: Start 2017-11-08 (Actual); Primary Completion 2020-03-18 (Actual); Study Completion 2020-04-08 (Actual)

PRIMARY OUTCOMES:
Relative risk of dengue in Wolbachia-treated versus untreated clusters | Up to 36 months participant enrolment
  Symptomatic, virologically-confirmed dengue virus (DENV) infection of any severity

SECONDARY OUTCOMES:
Relative risk of serotype-specific dengue in Wolbachia-treated versus untreated clusters | Up to 36 months participant enrolment
  Symptomatic, virologically-confirmed serotype-specific DENV infection of any severity.
Relative risk of Zika in Wolbachia-treated versus untreated clusters | Up to 36 months participant enrolment
  Symptomatic, virologically-confirmed Zika virus (ZIKV) infection of any severity.
Relative risk of Chikungunya in Wolbachia-treated versus untreated clusters | Up to 36 months participant enrolment
  Symptomatic, virologically-confirmed Chikungunya virus (CHIKV) infection of any severity.

CONTACTS AND LOCATIONS:
Overall Officials: Adi Utarini, MD, PhD, Principal Investigator — Faculty of Medicine, Universitas Gadjah Mada
Locations (1):
- Faculty of Medicine, Universitas Gadjah Mada, Yogyakarta, DIY, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Brady OJ, Gething PW, Bhatt S, Messina JP, Brownstein JS, Hoen AG, Moyes CL, Farlow AW, Scott TW, Hay SI. Refining the global spatial limits of dengue virus transmission by evidence-based consensus. PLoS Negl Trop Dis. 2012;6(8):e1760. doi: 10.1371/journal.pntd.0001760. Epub 2012 Aug 7. PMID 22880140
- [Background] Bhatt S, Gething PW, Brady OJ, Messina JP, Farlow AW, Moyes CL, Drake JM, Brownstein JS, Hoen AG, Sankoh O, Myers MF, George DB, Jaenisch T, Wint GR, Simmons CP, Scott TW, Farrar JJ, Hay SI. The global distribution and burden of dengue. Nature. 2013 Apr 25;496(7446):504-7. doi: 10.1038/nature12060. Epub 2013 Apr 7. PMID 23563266
- [Background] Shepard DS, Coudeville L, Halasa YA, Zambrano B, Dayan GH. Economic impact of dengue illness in the Americas. Am J Trop Med Hyg. 2011 Feb;84(2):200-7. doi: 10.4269/ajtmh.2011.10-0503. PMID 21292885
- [Background] Shepard DS, Undurraga EA, Halasa YA. Economic and disease burden of dengue in Southeast Asia. PLoS Negl Trop Dis. 2013;7(2):e2055. doi: 10.1371/journal.pntd.0002055. Epub 2013 Feb 21. PMID 23437406
- [Background] Shepard DS, Suaya JA, Halstead SB, Nathan MB, Gubler DJ, Mahoney RT, Wang DN, Meltzer MI. Cost-effectiveness of a pediatric dengue vaccine. Vaccine. 2004 Mar 12;22(9-10):1275-80. doi: 10.1016/j.vaccine.2003.09.019. PMID 15003657
- [Background] Dengue Vaccine Initiative. Dengue vaccine candidates in clinical development. (2016). Available at: http://www.denguevaccines.org/vaccine-development. (Accessed: 13th June 2016)
- [Background] L'Azou M, Moureau A, Sarti E, Nealon J, Zambrano B, Wartel TA, Villar L, Capeding MR, Ochiai RL; CYD14 Primary Study Group; CYD15 Primary Study Group. Symptomatic Dengue in Children in 10 Asian and Latin American Countries. N Engl J Med. 2016 Mar 24;374(12):1155-66. doi: 10.1056/NEJMoa1503877. PMID 27007959
- [Background] Capeding MR, Tran NH, Hadinegoro SR, Ismail HI, Chotpitayasunondh T, Chua MN, Luong CQ, Rusmil K, Wirawan DN, Nallusamy R, Pitisuttithum P, Thisyakorn U, Yoon IK, van der Vliet D, Langevin E, Laot T, Hutagalung Y, Frago C, Boaz M, Wartel TA, Tornieporth NG, Saville M, Bouckenooghe A; CYD14 Study Group. Clinical efficacy and safety of a novel tetravalent dengue vaccine in healthy children in Asia: a phase 3, randomised, observer-masked, placebo-controlled trial. Lancet. 2014 Oct 11;384(9951):1358-65. doi: 10.1016/S0140-6736(14)61060-6. Epub 2014 Jul 10. PMID 25018116
- [Background] Villar L, Dayan GH, Arredondo-Garcia JL, Rivera DM, Cunha R, Deseda C, Reynales H, Costa MS, Morales-Ramirez JO, Carrasquilla G, Rey LC, Dietze R, Luz K, Rivas E, Miranda Montoya MC, Cortes Supelano M, Zambrano B, Langevin E, Boaz M, Tornieporth N, Saville M, Noriega F; CYD15 Study Group. Efficacy of a tetravalent dengue vaccine in children in Latin America. N Engl J Med. 2015 Jan 8;372(2):113-23. doi: 10.1056/NEJMoa1411037. Epub 2014 Nov 3. PMID 25365753
- [Background] Guy B, Lang J, Saville M, Jackson N. Vaccination Against Dengue: Challenges and Current Developments. Annu Rev Med. 2016;67:387-404. doi: 10.1146/annurev-med-091014-090848. Epub 2015 Oct 23. PMID 26515983
- [Background] Hadinegoro SR, Arredondo-Garcia JL, Capeding MR, Deseda C, Chotpitayasunondh T, Dietze R, Muhammad Ismail HI, Reynales H, Limkittikul K, Rivera-Medina DM, Tran HN, Bouckenooghe A, Chansinghakul D, Cortes M, Fanouillere K, Forrat R, Frago C, Gailhardou S, Jackson N, Noriega F, Plennevaux E, Wartel TA, Zambrano B, Saville M; CYD-TDV Dengue Vaccine Working Group. Efficacy and Long-Term Safety of a Dengue Vaccine in Regions of Endemic Disease. N Engl J Med. 2015 Sep 24;373(13):1195-206. doi: 10.1056/NEJMoa1506223. Epub 2015 Jul 27. PMID 26214039
- [Background] Schilte C, Staikowsky F, Couderc T, Madec Y, Carpentier F, Kassab S, Albert ML, Lecuit M, Michault A. Chikungunya virus-associated long-term arthralgia: a 36-month prospective longitudinal study. PLoS Negl Trop Dis. 2013;7(3):e2137. doi: 10.1371/journal.pntd.0002137. Epub 2013 Mar 21. PMID 23556021
- [Background] Rolph MS, Foo SS, Mahalingam S. Emergent chikungunya virus and arthritis in the Americas. Lancet Infect Dis. 2015 Sep;15(9):1007-1008. doi: 10.1016/S1473-3099(15)00231-5. No abstract available. PMID 26333330
- [Background] Weaver SC, Costa F, Garcia-Blanco MA, Ko AI, Ribeiro GS, Saade G, Shi PY, Vasilakis N. Zika virus: History, emergence, biology, and prospects for control. Antiviral Res. 2016 Jun;130:69-80. doi: 10.1016/j.antiviral.2016.03.010. Epub 2016 Mar 18. PMID 26996139
- [Background] World Health Organization. Outcome of the Emergency Committee regarding clusters of microcephaly and Guillain-Barre syndrome. (2016)
- [Background] World Health Organization. Mosquito (vector) control emergency response and preparedness for Zika virus. (2016). Available at: http://www.who.int/neglected_diseases/news/mosquito_vector_control_response/en/. (Accessed: 18th March 2016)
- [Background] Karyanti MR, Uiterwaal CS, Kusriastuti R, Hadinegoro SR, Rovers MM, Heesterbeek H, Hoes AW, Bruijning-Verhagen P. The changing incidence of dengue haemorrhagic fever in Indonesia: a 45-year registry-based analysis. BMC Infect Dis. 2014 Jul 26;14:412. doi: 10.1186/1471-2334-14-412. PMID 25064368
- [Background] Graham RR, Juffrie M, Tan R, Hayes CG, Laksono I, Ma'roef C, Erlin, Sutaryo, Porter KR, Halstead SB. A prospective seroepidemiologic study on dengue in children four to nine years of age in Yogyakarta, Indonesia I. studies in 1995-1996. Am J Trop Med Hyg. 1999 Sep;61(3):412-9. doi: 10.4269/ajtmh.1999.61.412. PMID 10497982
- [Background] BPS - Statistics Indonesia. Badan Pusat Statistik. (2016). Available at: www.bps.go.id
- [Background] Ramadona AL, Lazuardi L, Hii YL, Holmner A, Kusnanto H, Rocklov J. Prediction of Dengue Outbreaks Based on Disease Surveillance and Meteorological Data. PLoS One. 2016 Mar 31;11(3):e0152688. doi: 10.1371/journal.pone.0152688. eCollection 2016. PMID 27031524
- [Background] Porter KR, Tan R, Istary Y, Suharyono W, Sutaryo, Widjaja S, Ma'Roef C, Listiyaningsih E, Kosasih H, Hueston L, McArdle J, Juffrie M. A serological study of Chikungunya virus transmission in Yogyakarta, Indonesia: evidence for the first outbreak since 1982. Southeast Asian J Trop Med Public Health. 2004 Jun;35(2):408-15. PMID 15691147
- [Background] Kosasih H, de Mast Q, Widjaja S, Sudjana P, Antonjaya U, Ma'roef C, Riswari SF, Porter KR, Burgess TH, Alisjahbana B, van der Ven A, Williams M. Evidence for endemic chikungunya virus infections in Bandung, Indonesia. PLoS Negl Trop Dis. 2013 Oct 24;7(10):e2483. doi: 10.1371/journal.pntd.0002483. eCollection 2013. PMID 24205417
- [Background] Riswari SF, Ma'roef CN, Djauhari H, Kosasih H, Perkasa A, Yudhaputri FA, Artika IM, Williams M, van der Ven A, Myint KS, Alisjahbana B, Ledermann JP, Powers AM, Jaya UA. Study of viremic profile in febrile specimens of chikungunya in Bandung, Indonesia. J Clin Virol. 2016 Jan;74:61-5. doi: 10.1016/j.jcv.2015.11.017. Epub 2015 Nov 17. PMID 26679829
- [Background] Laras K, Sukri NC, Larasati RP, Bangs MJ, Kosim R, Djauzi, Wandra T, Master J, Kosasih H, Hartati S, Beckett C, Sedyaningsih ER, Beecham HJ 3rd, Corwin AL. Tracking the re-emergence of epidemic chikungunya virus in Indonesia. Trans R Soc Trop Med Hyg. 2005 Feb;99(2):128-41. doi: 10.1016/j.trstmh.2004.03.013. PMID 15693148
- [Background] Mulyatno KC, Susilowati H, Yamanaka A, Soegijanto S, Konishi E. Primary isolation and phylogenetic studies of Chikungunya virus from Surabaya, Indonesia. Jpn J Infect Dis. 2012;65(1):92-4. No abstract available. PMID 22274167
- [Background] Haddow AD, Schuh AJ, Yasuda CY, Kasper MR, Heang V, Huy R, Guzman H, Tesh RB, Weaver SC. Genetic characterization of Zika virus strains: geographic expansion of the Asian lineage. PLoS Negl Trop Dis. 2012;6(2):e1477. doi: 10.1371/journal.pntd.0001477. Epub 2012 Feb 28. PMID 22389730
- [Background] Perkasa A, Yudhaputri F, Haryanto S, Hayati RF, Ma'roef CN, Antonjaya U, Yohan B, Myint KS, Ledermann JP, Rosenberg R, Powers AM, Sasmono RT. Isolation of Zika Virus from Febrile Patient, Indonesia. Emerg Infect Dis. 2016 May;22(5):924-5. doi: 10.3201/eid2205.151915. No abstract available. PMID 27088970
- [Background] Kwong JC, Druce JD, Leder K. Zika virus infection acquired during brief travel to Indonesia. Am J Trop Med Hyg. 2013 Sep;89(3):516-7. doi: 10.4269/ajtmh.13-0029. Epub 2013 Jul 22. PMID 23878182
- [Background] Leung GH, Baird RW, Druce J, Anstey NM. ZIKA VIRUS INFECTION IN AUSTRALIA FOLLOWING A MONKEY BITE IN INDONESIA. Southeast Asian J Trop Med Public Health. 2015 May;46(3):460-4. PMID 26521519
- [Background] Esu E, Lenhart A, Smith L, Horstick O. Effectiveness of peridomestic space spraying with insecticide on dengue transmission; systematic review. Trop Med Int Health. 2010 May;15(5):619-31. doi: 10.1111/j.1365-3156.2010.02489.x. Epub 2010 Mar 8. PMID 20214764
- [Background] Pilger, D., De Maesschalck, M., Horstick, O. & San Martín, J. L. Dengue outbreak response: documented effective interventions and evidence gaps. TropIKA 1, (2010)
- [Background] Erlanger TE, Keiser J, Utzinger J. Effect of dengue vector control interventions on entomological parameters in developing countries: a systematic review and meta-analysis. Med Vet Entomol. 2008 Sep;22(3):203-21. doi: 10.1111/j.1365-2915.2008.00740.x. PMID 18816269
- [Background] Bowman LR, Runge-Ranzinger S, McCall PJ. Assessing the relationship between vector indices and dengue transmission: a systematic review of the evidence. PLoS Negl Trop Dis. 2014 May 8;8(5):e2848. doi: 10.1371/journal.pntd.0002848. eCollection 2014 May. PMID 24810901
- [Background] Bowman LR, Donegan S, McCall PJ. Is Dengue Vector Control Deficient in Effectiveness or Evidence?: Systematic Review and Meta-analysis. PLoS Negl Trop Dis. 2016 Mar 17;10(3):e0004551. doi: 10.1371/journal.pntd.0004551. eCollection 2016 Mar. PMID 26986468
- [Background] Andersson N, Nava-Aguilera E, Arostegui J, Morales-Perez A, Suazo-Laguna H, Legorreta-Soberanis J, Hernandez-Alvarez C, Fernandez-Salas I, Paredes-Solis S, Balmaseda A, Cortes-Guzman AJ, Serrano de Los Santos R, Coloma J, Ledogar RJ, Harris E. Evidence based community mobilization for dengue prevention in Nicaragua and Mexico (Camino Verde, the Green Way): cluster randomized controlled trial. BMJ. 2015 Jul 8;351:h3267. doi: 10.1136/bmj.h3267. PMID 26156323
- [Background] Degener CM, Eiras AE, Azara TM, Roque RA, Rosner S, Codeco CT, Nobre AA, Rocha ES, Kroon EG, Ohly JJ, Geier M. Evaluation of the effectiveness of mass trapping with BG-sentinel traps for dengue vector control: a cluster randomized controlled trial in Manaus, Brazil. J Med Entomol. 2014 Mar;51(2):408-20. doi: 10.1603/me13107. PMID 24724291
- [Background] Wilson AL, Boelaert M, Kleinschmidt I, Pinder M, Scott TW, Tusting LS, Lindsay SW. Evidence-based vector control? Improving the quality of vector control trials. Trends Parasitol. 2015 Aug;31(8):380-90. doi: 10.1016/j.pt.2015.04.015. Epub 2015 May 19. PMID 25999026
- [Background] O'Neill SL, Pettigrew MM, Sinkins SP, Braig HR, Andreadis TG, Tesh RB. In vitro cultivation of Wolbachia pipientis in an Aedes albopictus cell line. Insect Mol Biol. 1997 Feb;6(1):33-9. doi: 10.1046/j.1365-2583.1997.00157.x. PMID 9013253
- [Background] Stouthamer R, Breeuwer JA, Hurst GD. Wolbachia pipientis: microbial manipulator of arthropod reproduction. Annu Rev Microbiol. 1999;53:71-102. doi: 10.1146/annurev.micro.53.1.71. PMID 10547686
- [Background] Rousset F, Vautrin D, Solignac M. Molecular identification of Wolbachia, the agent of cytoplasmic incompatibility in Drosophila simulans, and variability in relation with host mitochondrial types. Proc Biol Sci. 1992 Mar 23;247(1320):163-8. doi: 10.1098/rspb.1992.0023. PMID 1350096
- [Background] Hilgenboecker K, Hammerstein P, Schlattmann P, Telschow A, Werren JH. How many species are infected with Wolbachia?--A statistical analysis of current data. FEMS Microbiol Lett. 2008 Apr;281(2):215-20. doi: 10.1111/j.1574-6968.2008.01110.x. Epub 2008 Feb 28. PMID 18312577
- [Background] McMeniman CJ, Lane RV, Cass BN, Fong AW, Sidhu M, Wang YF, O'Neill SL. Stable introduction of a life-shortening Wolbachia infection into the mosquito Aedes aegypti. Science. 2009 Jan 2;323(5910):141-4. doi: 10.1126/science.1165326. PMID 19119237
- [Background] Joubert DA, Walker T, Carrington LB, De Bruyne JT, Kien DH, Hoang Nle T, Chau NV, Iturbe-Ormaetxe I, Simmons CP, O'Neill SL. Establishment of a Wolbachia Superinfection in Aedes aegypti Mosquitoes as a Potential Approach for Future Resistance Management. PLoS Pathog. 2016 Feb 18;12(2):e1005434. doi: 10.1371/journal.ppat.1005434. eCollection 2016 Feb. PMID 26891349
- [Background] Walker T, Johnson PH, Moreira LA, Iturbe-Ormaetxe I, Frentiu FD, McMeniman CJ, Leong YS, Dong Y, Axford J, Kriesner P, Lloyd AL, Ritchie SA, O'Neill SL, Hoffmann AA. The wMel Wolbachia strain blocks dengue and invades caged Aedes aegypti populations. Nature. 2011 Aug 24;476(7361):450-3. doi: 10.1038/nature10355. PMID 21866159
- [Background] Dutra HL, Rocha MN, Dias FB, Mansur SB, Caragata EP, Moreira LA. Wolbachia Blocks Currently Circulating Zika Virus Isolates in Brazilian Aedes aegypti Mosquitoes. Cell Host Microbe. 2016 Jun 8;19(6):771-4. doi: 10.1016/j.chom.2016.04.021. Epub 2016 May 4. PMID 27156023
- [Background] Johnson KN. The Impact of Wolbachia on Virus Infection in Mosquitoes. Viruses. 2015 Nov 4;7(11):5705-17. doi: 10.3390/v7112903. PMID 26556361
- [Background] Rainey SM, Shah P, Kohl A, Dietrich I. Understanding the Wolbachia-mediated inhibition of arboviruses in mosquitoes: progress and challenges. J Gen Virol. 2014 Mar;95(Pt 3):517-530. doi: 10.1099/vir.0.057422-0. Epub 2013 Dec 16. PMID 24343914
- [Background] Amuzu HE, Simmons CP, McGraw EA. Effect of repeat human blood feeding on Wolbachia density and dengue virus infection in Aedes aegypti. Parasit Vectors. 2015 Apr 24;8:246. doi: 10.1186/s13071-015-0853-y. PMID 25903749
- [Background] Ye YH, Carrasco AM, Frentiu FD, Chenoweth SF, Beebe NW, van den Hurk AF, Simmons CP, O'Neill SL, McGraw EA. Wolbachia Reduces the Transmission Potential of Dengue-Infected Aedes aegypti. PLoS Negl Trop Dis. 2015 Jun 26;9(6):e0003894. doi: 10.1371/journal.pntd.0003894. eCollection 2015. PMID 26115104
- [Background] Frentiu FD, Zakir T, Walker T, Popovici J, Pyke AT, van den Hurk A, McGraw EA, O'Neill SL. Limited dengue virus replication in field-collected Aedes aegypti mosquitoes infected with Wolbachia. PLoS Negl Trop Dis. 2014 Feb 20;8(2):e2688. doi: 10.1371/journal.pntd.0002688. eCollection 2014 Feb. PMID 24587459
- [Background] Moreira LA, Iturbe-Ormaetxe I, Jeffery JA, Lu G, Pyke AT, Hedges LM, Rocha BC, Hall-Mendelin S, Day A, Riegler M, Hugo LE, Johnson KN, Kay BH, McGraw EA, van den Hurk AF, Ryan PA, O'Neill SL. A Wolbachia symbiont in Aedes aegypti limits infection with dengue, Chikungunya, and Plasmodium. Cell. 2009 Dec 24;139(7):1268-78. doi: 10.1016/j.cell.2009.11.042. PMID 20064373
- [Background] Ferguson NM, Kien DT, Clapham H, Aguas R, Trung VT, Chau TN, Popovici J, Ryan PA, O'Neill SL, McGraw EA, Long VT, Dui le T, Nguyen HL, Chau NV, Wills B, Simmons CP. Modeling the impact on virus transmission of Wolbachia-mediated blocking of dengue virus infection of Aedes aegypti. Sci Transl Med. 2015 Mar 18;7(279):279ra37. doi: 10.1126/scitranslmed.3010370. PMID 25787763
- [Background] Wolbers M, Kleinschmidt I, Simmons CP, Donnelly CA. Considerations in the design of clinical trials to test novel entomological approaches to dengue control. PLoS Negl Trop Dis. 2012;6(11):e1937. doi: 10.1371/journal.pntd.0001937. Epub 2012 Nov 29. No abstract available. PMID 23209869
- [Background] Hayes, R. & Moulton, L. Cluster randomized trials. (Chapman & Hall/CRC, 2009)
- [Background] Endy TP, Yoon IK, Mammen MP. Prospective cohort studies of dengue viral transmission and severity of disease. Curr Top Microbiol Immunol. 2010;338:1-13. doi: 10.1007/978-3-642-02215-9_1. PMID 19802574
- [Background] Vandenbroucke JP, Pearce N. Case-control studies: basic concepts. Int J Epidemiol. 2012 Oct;41(5):1480-9. doi: 10.1093/ije/dys147. PMID 23045208
- [Background] De Serres G, Skowronski DM, Wu XW, Ambrose CS. The test-negative design: validity, accuracy and precision of vaccine efficacy estimates compared to the gold standard of randomised placebo-controlled clinical trials. Euro Surveill. 2013 Sep 12;18(37):20585. doi: 10.2807/1560-7917.es2013.18.37.20585. PMID 24079398
- [Background] Greenland S, Thomas DC. On the need for the rare disease assumption in case-control studies. Am J Epidemiol. 1982 Sep;116(3):547-53. doi: 10.1093/oxfordjournals.aje.a113439. PMID 7124721
- [Background] Jackson ML, Nelson JC. The test-negative design for estimating influenza vaccine effectiveness. Vaccine. 2013 Apr 19;31(17):2165-8. doi: 10.1016/j.vaccine.2013.02.053. Epub 2013 Mar 13. PMID 23499601
- [Background] Haber M, An Q, Foppa IM, Shay DK, Ferdinands JM, Orenstein WA. A probability model for evaluating the bias and precision of influenza vaccine effectiveness estimates from case-control studies. Epidemiol Infect. 2015 May;143(7):1417-26. doi: 10.1017/S0950268814002179. Epub 2014 Aug 22. PMID 25147970
- [Background] Smith PG, Morrow RH, Ross DA, editors. Field Trials of Health Interventions: A Toolbox. 3rd edition. Oxford (UK): OUP Oxford; 2015 Jun 1. Available from http://www.ncbi.nlm.nih.gov/books/NBK305515/ PMID 26225404
- [Background] Ivers NM, Halperin IJ, Barnsley J, Grimshaw JM, Shah BR, Tu K, Upshur R, Zwarenstein M. Allocation techniques for balance at baseline in cluster randomized trials: a methodological review. Trials. 2012 Aug 1;13:120. doi: 10.1186/1745-6215-13-120. PMID 22853820
- [Background] Haybittle JL. Repeated assessment of results in clinical trials of cancer treatment. Br J Radiol. 1971 Oct;44(526):793-7. doi: 10.1259/0007-1285-44-526-793. No abstract available. PMID 4940475
- [Derived] Utarini A, Indriani C, Ahmad RA, Tantowijoyo W, Arguni E, Ansari MR, Supriyati E, Wardana DS, Meitika Y, Ernesia I, Nurhayati I, Prabowo E, Andari B, Green BR, Hodgson L, Cutcher Z, Rances E, Ryan PA, O'Neill SL, Dufault SM, Tanamas SK, Jewell NP, Anders KL, Simmons CP; AWED Study Group. Efficacy of Wolbachia-Infected Mosquito Deployments for the Control of Dengue. N Engl J Med. 2021 Jun 10;384(23):2177-2186. doi: 10.1056/NEJMoa2030243. PMID 34107180
- [Derived] Anders KL, Indriani C, Ahmad RA, Tantowijoyo W, Arguni E, Andari B, Jewell NP, Dufault SM, Ryan PA, Tanamas SK, Rances E, O'Neill SL, Simmons CP, Utarini A. Update to the AWED (Applying Wolbachia to Eliminate Dengue) trial study protocol: a cluster randomised controlled trial in Yogyakarta, Indonesia. Trials. 2020 May 25;21(1):429. doi: 10.1186/s13063-020-04367-2. PMID 32450914
- [Derived] Anders KL, Indriani C, Ahmad RA, Tantowijoyo W, Arguni E, Andari B, Jewell NP, Rances E, O'Neill SL, Simmons CP, Utarini A. The AWED trial (Applying Wolbachia to Eliminate Dengue) to assess the efficacy of Wolbachia-infected mosquito deployments to reduce dengue incidence in Yogyakarta, Indonesia: study protocol for a cluster randomised controlled trial. Trials. 2018 May 31;19(1):302. doi: 10.1186/s13063-018-2670-z. PMID 29855331

DOCUMENTS (1):
  • Statistical Analysis Plan (2020-05-28): https://cdn.clinicaltrials.gov/large-docs/85/NCT03055585/SAP_002.pdf